CLINICAL TRIAL: NCT01664130
Title: High-Dose Stereotactic Body Radiation Therapy in Treating Patients With Low-, Intermediate-, or High-Risk Localized Prostate Cancer
Brief Title: High-Dose Stereotactic Radiation for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1812; NCI-2012-01252 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (SBRT) (Experimental): Patients undergo 5 fractions of prostate stereotactic body radiation therapy over 10-20 days with at least 40 hours between each fraction in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: stereotactic body radiation therapy; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies high-dose stereotactic body radiation therapy (SBRT) in treating patients with low-, intermediate-, or high-risk localized prostate cancer. SBRT may be able to send x-rays directly to the tumor and cause less damage to normal tissue

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess treatment related gastrointestinal (GI) and genitourinary (GU) toxicity for patients who undergo SBRT for localized prostate cancer.

SECONDARY OBJECTIVES:

I. Follow quality of life after SBRT using Expanded Prostate Cancer Index Composite (EPIC) and American Urological Association (AUA) scores.

II. Assess biochemical control after high-dose SBRT.

OUTLINE:

Patients undergo 5 fractions of prostate stereotactic body radiation therapy over 10-12 days with at least 40 hours between each fraction in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1.5, 4, 8, and 12 months, every 6 months for 4 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have prostate adenocarcinoma proven by histologic diagnosis
* The patient must have clinical stage T1a-T3b with localized prostate cancer considered low, intermediate, or high risk as defined by the National Comprehensive Cancer Network (NCCN) guidelines; any patient whom is defined as high-risk must undergo screening with computed tomography (CT) or magnetic resonance imaging (MRI) of the abdomen and pelvis as well as bone scan prior to enrollment for staging purposes; low and intermediate risk patients do not require imaging for staging unless they have a focal symptom warranting investigation
* Performance status - Karnofsky performance status (PS) >= 70
* Life expectancy of > 5 years, in the opinion of and as documented by the investigator
* Patients must either already have fiducials already placed within the prostate, or otherwise be candidates for prostate fiducial placement (no bleeding disorders which may cause excessive bleeding with fiducial placement, INR < 2.0).
* Patients must have prostate-specific antigen (PSA) drawn within the 90 days prior to enrollment
* Men must agree to use adequate contraception (double barrier method of birth control or abstinence) for the duration of study participation and for 12 months after completing treatment
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior treatment toxicities must be resolved to =< grade 1 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
* Patients who are receiving any other investigational agents
* Evidence of metastatic disease prior to radiation
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Prior pelvic radiation therapy
* Patients whom are planned to receive pelvic nodal radiation are excluded
* Weight > 350 lbs
* Contraindications to placement of fiducials required for high-precision image guidance (e.g. bleeding disorders which may cause excessive bleeding with placement, requirement for coumadin, international normalized ratio [INR] > 2.0)
* Patients unable to maintain a full bladder during treatment
* Previous prostatectomy
* Inflammatory bowel disease
* AUA score > 15 in spite of optimal therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Stephans, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Parsai S, Juloori A, Sedor G, Reddy CA, Thousand R, Magnelli A, Berglund RK, Stovsky M, Klein EA, Tendulkar RD, Stephans KL. Heterogenous Dose-escalated Prostate Stereotactic Body Radiation Therapy for All Risk Prostate Cancer: Quality of Life and Clinical Outcomes of an Institutional Pilot Study. Am J Clin Oncol. 2020 Jul;43(7):469-476. doi: 10.1097/COC.0000000000000693. PMID 32349020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from regional hospitals from July 2012 thru Jan 2015.
Period: Overall Study
Arm/Group | Treatment (SBRT)
Started | 35
Completed | 33
Not Completed | 2
Not completed — competing secondary disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 35
Age, Customized [Count of Participants; unit: Participants]
  50-59 yrs | 6
  60-69 yrs | 12
  70-79 yrs | 15
  80-89 yrs | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Related GI and/or GU Toxicity as Assessed by the NCI CTCTAE Version 4.0
Description: Number of patients with excessive GI and/or GU toxicity, defined as a grade 3 GU toxicity rate of ≥15% according to the NCI CTCTAE version 4.0
Time Frame: 1.5 months
Population: All patients that received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 35
Participants | 1

2. Primary Outcome: Number of Patients With Treatment Related GI and GU Toxicity as Assessed by the NCI CTCTAE Version 4.0
Description: as for outcome 1
Time Frame: 4 months
Population: Per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 35
Participants | 0

3. Primary Outcome: Number of Patients With Treatment Related GI and GU Toxicity as Assessed by the NCI CTCTAE Version 4.0
Description: as for outcome 1
Time Frame: 8 months
Population: Per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 35
Participants | 0

4. Primary Outcome: Number of Patients With Treatment Related GI and GU Toxicity as Assessed by the NCI CTCTAE Version 4.0
Description: as for outcome 1
Time Frame: 12 months
Population: All patients that received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 35
Participants | 0

5. Secondary Outcome: Quality of Life as Assessed by EPIC Scores
Description: Quality of life (QOL) from baseline as assessed by scores of the EPIC Questionnaire. Scores for each domain (urinary incontinence, bowel, sexual, hormonal) range from 0-100, with higher scores indicating better clinical assessment.
Time Frame: Baseline and 1.5 months
Population: Participants that were able to complete the questionnaire at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Before treatment
- After Treatment (SBRT): After treatment (SBRT)
  Patients undergo 5 fractions of prostate stereotactic body radiation therapy over 10-20 days with at least 40 hours between each fraction in the absence of disease progression or unacceptable toxicity.
  stereotactic body radiation therapy: Undergo SBRT
  quality-of-life assessment: Ancillary studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Baseline | After Treatment (SBRT)
Number analyzed (Participants) | 31 | 32
score on a scale
  Urinary Incontenence Domain | 83.2 (16.5) | 84.0 (18.7)
  Bowel Domain | 90.5 (12.4) | 83.7 (22.7)
  Sexual Function Domain | 46.4 (30.4) | 36.8 (28.3)
  Hormonal Domain | 80.6 (19.4) | 76.6 (20.7)

6. Secondary Outcome: Quality of Life as Assessed by EPIC Scores
Description: as for outcome 5
Time Frame: Baseline and 4 months
Population: Participants that were able to complete the questionnaire at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | After Treatment (SBRT)
Number analyzed (Participants) | 32 | 33
score on a scale
  Urinary Incontenence Domain | 83.2 (16.5) | 85.0 (16.3)
  Bowel Domain | 90.5 (12.4) | 85.6 (21.1)
  Sexual Function Domain | 46.4 (30.4) | 33.6 (31.1)
  Hormonal Domain | 80.6 (19.4) | 79.4 (22.6)

7. Secondary Outcome: Quality of Life as Assessed by EPIC Scores
Description: as for outcome 5
Time Frame: Baseline and 8 months
Population: Participants that were able to complete the questionnaire at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | After Treatment (SBRT)
Number analyzed (Participants) | 31 | 32
score on a scale
  Urinary Incontenence Domain | 83.2 (16.5) | 85.7 (17.3)
  Bowel Domain | 90.5 (12.4) | 86.6 (19.3)
  Sexual Function Domain | 46.4 (30.4) | 37.5 (29.0)
  Hormonal Domain | 80.6 (19.4) | 82.4 (16.7)

8. Secondary Outcome: Quality of Life as Assessed by EPIC Scores
Description: as for outcome 5
Time Frame: Baseline and 12 months
Population: Participants that were able to complete the questionnaire at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | After Treatment (SBRT)
Number analyzed (Participants) | 31 | 34
score on a scale
  Urinary Incontenence Domain | 83.2 (16.5) | 83.4 (19.4)
  Bowel Domain | 90.5 (12.4) | 86.3 (18.4)
  Sexual Function Domain | 46.4 (30.4) | 37.1 (28.5)
  Hormonal Domain | 80.6 (19.4) | 87.3 (12.3)

9. Secondary Outcome: Quality of Life as Assessed by Change in AUA Scores
Description: Quality of life (QOL) as assessed by changes in AUA scores ranging between 0 to 35, with higher scores indicating a worse clinical assessment.
Time Frame: Baseline and 1.5 months
Population: Participants that were able to complete the questionnaire at specific time point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 32
score on a scale | 9 [1 to 25]

10. Secondary Outcome: Quality of Life as Assessed by Change in AUA Scores
Description: as for outcome 9
Time Frame: Baseline and 4 months
Population: Participants that were able to complete the questionnaire at specific time point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 32
score on a scale | 7.5 [0 to 29]

11. Secondary Outcome: Quality of Life as Assessed by Change in AUA Scores
Description: as for outcome 9
Time Frame: Baseline and 8 months
Population: Participants that were able to complete the questionnaire at specific time point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 31
score on a scale | 6 [0 to 21]

12. Secondary Outcome: Quality of Life as Assessed by Change in AUA Scores
Description: as for outcome 9
Time Frame: Baseline and 12 months
Population: Participants that were able to complete the questionnaire at specific time point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 33
score on a scale | 8 [0 to 33]

13. Secondary Outcome: Percentage of Participants With Biochemical Relapse Free Survival as Measured by Serum PSA
Description: Percentage of Participants with biochemical failure. Biochemical failure is defined as a rise in PSA of 2.0 ng/dl above the post-treatment nadir.
Time Frame: Baseline and 1.5 months
Population: participants who had a PSA values up to the reporting time interval. Not every patient had all of the PSA values collected due to missed test visits.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 29
percentage of participants | 100 [100 to 100]

14. Secondary Outcome: Percentage of Participants With Biochemical Relapse Free Survival as Measured by Serum PSA
Description: Biochemical failure will be defined as a rise in PSA of 2.0 ng/dl above the post-treatment nadir.
Time Frame: Baseline and 4 months
Population: participants who had a PSA value up to the reporting time interval. Not every patient had all of the PSA values collected due to missed test visits.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 29
percentage of participants | 100 [100 to 100]

15. Secondary Outcome: Percentage of Participants With Biochemical Relapse Free Survival as Measured by Serum PSA
Description: Biochemical failure will be defined as a rise in PSA of 2.0 ng/dl above the post-treatment nadir.
Time Frame: Baseline and 8 months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 27
percentage of participants | 96.5 [89.7 to 100]

16. Secondary Outcome: Percentage of Participants With Biochemical Relapse Free Survival as Measured by Serum PSA
Description: Percent measurement of biochemical failure will be defined as a rise in PSA of 2.0 ng/dl above the post-treatment nadir.
Time Frame: Baseline and 12 months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 27
percentage of participants | 96.5 [89.7 to 100]

ADVERSE EVENTS:
Time Frame: Adverse event data collect from participants up to 1 year in follow-up.
Arm/Group | Treatment (SBRT)
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SBRT) (N=35)
Prostate infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SBRT) (N=35)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Fatigue (General disorders) | 15 (16)
Hematuria (Renal and urinary disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 6 (7)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 18 (22)
Urinary incontinence (Renal and urinary disorders) | 7 (7)
Urinary retention (Renal and urinary disorders) | 13 (14)
Urinary tract pain (Renal and urinary disorders) | 7 (9)
Urinary urgency (Renal and urinary disorders) | 14 (17)
Weight gain (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes